CLINICAL TRIAL: NCT02235779
Title: DIagnostic Yield of Transbronchial Cryobiopsies in Subjects With Interstitial Lung Disease
Brief Title: Diagnostic Yield of Transbronchial Cryobiopsy in Diagnosis of Interstitial Lung Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CryobiopsieTBB
Record Dates: First submitted 2014-08-26; First posted 2014-09-10 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Interstitial Lung Disease
Keywords: ILD; Pulmonary fibrosis; Cryobiopsy; Transbronchial
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryobiopsy (Other)
  Interventions: Other: Transbronchial lung cryobiopsy

INTERVENTIONS:
Other: Transbronchial lung cryobiopsy

SUMMARY:
Evaluation of diagnostic yield, feasibility and safety of transbronchial lung cryobiopsies done via bronchoscopy in the investigation of interstitial lung disease in comparison with videothoracoscopy-assisted surgical lung biopsy.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subjects with interstitial lung disease in whom a surgical lung biopsy is planned for diagnostic investigation.

Exclusion Criteria:

* Aged less than 18 y.o.
* Pregnancy
* Known coagulatoin disorder or blood dyscrasia
* Aaking antiplatelet agents other than aspirin or therapeutic anticoagulants drugs that cannot be safely discontinued to undergo lung biopsy
* Arterial oxgen pressure less than 60 mmHg on more than 2 liters per minute oxygen
* Known pulmonary hypertension defined as systolic PAP above 40 mmHg on echocardiography
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-08; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall diagnostic yield of cryobiopsy specimens in interstitial lung disease | After biopsy (up to 24 months)
  Number of cryobiopsy specimens from which a specific diagnosis of interstitial lung disease can be ascertained, as assessed by a two different pathologists blinded to the known final diagnosis.

SECONDARY OUTCOMES:
Complication rate of transbronchial cryobiopsy procedure | Per-procedure and up to 24 hours after
  Assessment of complications related to cryoTBB:
  * pneumothorax
  * hemorrage
  * other complications
Number of diagnostic specimens of cryoTBB in comparison with surgical lung biopsy specimen | After biopsy (up to 24 months)
  Diagnostic concordance between cryobiopsy specimen analysis and corresponding surgical lung biopsy done in same subjects (same lung/lobe)
Inter-observer agreement for cryobiopsy specimens | After biopsy (up to 24 months)
  Interobserver agreement rate between two different pathologists blinded to subject history/radiological record and surgical lung biopsy specimen.
Size of cryobiopsy specimen | After biopsy (up to 24months)
  Size of TBB cryobiopsy specimen measured by two different pathologists responsible for its interpretation.
Quality of cyrobiopsy specimens | After biopsy (up to 24 months)
  Pathological quality score of TBB cryobiopsy specimens (artefacts, size, etc.) as assessed by two different pathologists responsible for their interpretation.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Delage, MDCM, Study Chair — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

REFERENCES:
- [Derived] Fortin M, Liberman M, Delage A, Dion G, Martel S, Rolland F, Soumagne T, Trahan S, Assayag D, Albert E, Kelly MM, Johannson KA, Guenther Z, Leduc C, Manganas H, Prenovault J, Provencher S. Transbronchial Lung Cryobiopsy and Surgical Lung Biopsy: A Prospective Multi-Centre Agreement Clinical Trial (CAN-ICE). Am J Respir Crit Care Med. 2023 Jun 15;207(12):1612-1619. doi: 10.1164/rccm.202209-1812OC. PMID 36796092